CLINICAL TRIAL: NCT03743974
Title: Analgesic Efficacy of Ultrasound-Guided Interscalene Block Versus Supraclavicular Block for Ambulatory Arthroscopic Rotator Cuff Repair: a Prospective, Randomized, Single-blind, Comparative Study
Brief Title: Analgesic Efficacy of US-Guided Interscalene Block Versus Supraclavicular Block for Ambulatory Arthroscopic Rotator Cuff Repair
Acronym: BISBSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Hôpital Privé Jean Mermoz. Service Dr Julien Cabaton (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGDS BISBSC
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Shoulder Lesions
Keywords: arthroscopic shoulder surgery; interscalene block analgesia; supraclavicular block analgesia; Ambulatory surgery for rotator cuff
MeSH Terms: interventions — Placental Lactogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene block (Active Comparator): Site of injection for ISB was the C6 plexus nerve root with a posterior in-plane approach, with neurostimulation control, and ultrasound-controlled of extra-plexus injection of the mixture posterior to the C6 root
  Interventions: Procedure: arthroscopic shoulder surgery of rotary cuff (ISB)
- Supraclavicular block (Experimental): Site of injection for SCB was superficial and lateral to the trunks of the brachial plexus, and not directly deep inside the "corner pocket" zone, with neurostimulation control and visualization of the lung
  Interventions: Procedure: arthroscopic shoulder surgery of rotary cuff (CSB)

INTERVENTIONS:
Procedure: arthroscopic shoulder surgery of rotary cuff (ISB) — ISB were performed in the same manner by one of the two anesthesiologists in our team: (i) patients were monitored, after sedation with sublingual midazolam (0.1 mg/kg) + a single bolus of intravenous (IV) ketamine (0.2 mg/kg); (ii) ultrasound-guidance was carried out using a Kontron® or General Electric® ultrasound machine; (iii) neurostimulation was performed with a Stimuplex HNS® 12 set at 0.1 ms, 1 Hz and 1 mA stimulation, in sentinel mode, with the aim of securing the approach of the needle; (iv) a single perineural injection was performed with a 50 mm Vygon® needle containing a mixture of 100 mg levobupivacaine (20 mL, 0.5%) and clonidine (1 µg/kg patient) as is the local common protocol and in the absence of contraindications.
  Arms: Interscalene block
Procedure: arthroscopic shoulder surgery of rotary cuff (CSB) — SCB were performed in the same manner by one of the two anesthesiologists in our team: (i) patients were monitored, after sedation with sublingual midazolam (0.1 mg/kg) + a single bolus of intravenous (IV) ketamine (0.2 mg/kg); (ii) ultrasound-guidance was carried out using a Kontron® or General Electric® ultrasound machine; (iii) neurostimulation was performed with a Stimuplex HNS® 12 set at 0.1 ms, 1 Hz and 1 mA stimulation, in sentinel mode, with the aim of securing the approach of the needle; (iv) a single perineural injection was performed with a 50 mm Vygon® needle containing a mixture of 100 mg levobupivacaine (20 mL, 0.5%) and clonidine (1 µg/kg patient) as is the local common protocol and in the absence of contraindications.
  Arms: Supraclavicular block

SUMMARY:
Ultrasound-guided interscalene block (ISB) is the reference technique for pain control after ambulatory upper limb surgery, but supraclavicular block (SCB) is an alternative procedure. We compared the efficacy of these two techniques in patients undergoing ambulatory arthroscopic rotator cuff repair (ARCR).

DETAILED DESCRIPTION:
The number of patients undergoing ambulatory arthroscopic rotator cuff repair (ARCR) in our center is increasing annually. This procedure is associated with significant postoperative pain and effective analgesia is required in order to develop day-case surgery. Although continuous interscalene catheter block (ISB) is considered to be the most effective analgesic technique for ARCR, the difficulties in implementing and monitoring ISB have led to many anesthesiologists preferring single injection block, so that patients can be discharged on the same day as surgery with a satisfactory level of pain control.

ISB is frequently associated with phrenic nerve block,even with low volumes of local anesthetics. Phrenic nerve block is a concern in some ambulatory surgery patients as it may lead to respiratory complications after hospital discharge, limiting the eligibility of many patients for day surgery. Changes in spirometry variables have been associated with ISB, whatever the site of injection around the roots (anterior or posterior). Nevertheless, effective regional anesthesia (RA) is essential for this surgery, because multimodal analgesia alone is insufficient.

Several alternatives to ISB exist that are associated with a decreased prevalence of phrenic nerve paresis.6 Supraclavicular block (SCB) decreases the risk of phrenic nerve involvement, particularly when guided by ultrasound. This technique, which has been linked to a risk of pneumothorax when carried out by neurostimulation only, has now been revived and is included among the RA techniques considered to be safe in terms of respiratory risk, especially when guided by ultrasound. Many studies have demonstrated a decreased risk of phrenic paresis with ultrasound-guided SCB, even with volumes as high as 20 mL. Published studies have demonstrated that SCB is an effective alternative to ISB, and many studies have shown that ultrasound-guided SCB is a safe technique for ambulatory shoulder surgery in terms of respiratory complications. SCB is therefore a real alternative to ISB for ambulatory ARCR, but comparative studies are necessary to evaluate its analgesic efficacy after patients have been discharged from hospital, particularly in terms of their oral morphine consumption at home.

Investigators carried out a monocentric, prospective, comparative study to determine whether SCB is non-inferior to ISB in terms of post-operative analgesia in patients undergoing ambulatory ARCR. Analgesic efficacy was determined by oral morphine use and/or pain scores in patients after hospital discharge. Promotor hypothesis was that SCB would provide similar or better analgesia to ISB in patients returning home on the evening of their surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patients were adults undergoing ARCR by a single surgeon (NJ), under RA and general anesthesia (GA);
* Returning home on the evening of their surgery (hospital stay <12 h);
* Patients adults ;
* Patients with social health insurance ;
* Patient able to understand the objective and constrains of the study.

Exclusion criteria:

* patients enable to return home on the evening of their surgery (for a medical or other reason);
* patients taking oral morphine derivatives before their surgery;
* patients with a contraindication for RA or in whom RA was not performed; those with a contraindication for oral morphine derivatives;
* patients who developed a complication during implementation of RA;
* patients refusing to participate in the study;
* patients whose consent was not recorded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
non-inferiority of BSC in relation to BIS on postoperative analgesic efficacy for arthroscopic outpatient shoulder rotator cuff repair surgery. | 2 days
  Opioid oral consumption at home within 48 hours of returning home.

IPD SHARING:
Plan to Share IPD: No